CLINICAL TRIAL: NCT05999396
Title: First in Human Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Efficacy of the Bispecific CD276xCD3 Antibody CC-3 in Patients With Colorectal Cancer
Brief Title: FIH, Bispecific CD276xCD3 Antibody CC-3 in Patients With Colorectal Cancer
Acronym: CoRe_CC-3
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CoRe_CC-3
Record Dates: First submitted 2023-07-20; First posted 2023-08-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Breast Carcinoma; Sarcoma; Penile Carcinoma
Keywords: new therapy; bispecific antibody; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Sarcoma; Penile Neoplasms

STUDY DESIGN:
Intervention Model Description: Open-label, multicenter, dose escalation and dose expansion part, Phase I clinical trial, designed to gain evidence of maximally tolerated and recommended phase-II dose of CC-3 in adult patients with CRC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of CC-3, a bispecific CD276xCD3 antibody (Experimental): The DL in the accelerated titration phase is fixed in each patient and is applied once per week. The start dose for the first patient is 20µg. Dose increase in the next patient is determined by SRC, comprised of investigators and Sponsor, and can be up to 100% based on safety, PK and PD data. Accelerated titration is terminated and switched to a standard 3 + 3 design in case of any AE Grade ≥ 2 (except AEs unequivocally due to underlying disease or an extraneous cause), occurrence of DLT or decision of SRC based on PK, PD, and safety data.
  In the dose expansion part, additional patients are treated to have 20 evaluabale patients at the MTD level defined in the dose escalation part.
  Interventions: Drug: Administration of CC-3

INTERVENTIONS:
Drug: Administration of CC-3 — Accelerated titration phase, Standard 3+3 titration phase, expansion phase

SUMMARY:
This trial is a first in human (FIH) clinical trial in patients with Colorectal cancer (CRC) after failure of at least three lines of previous therapy aiming to evaluate safety and efficacy of CC-3, a bispecific antibody (bsAb) with CD276xCD3 specificity developed within DKTK. CC-3 binds to CD276 on cancer cells as well as to tumor vessels of CRC, thereby allowing for a dual mode of anti-cancer action. CC-3 was developed in a novel format which not only prolongs serum half-life, but most importantly reduces off-target T cell activation with expected fewer side effects. A similar construct in this format with PSMAxCD3 specificity is presently undergoing clinical evaluation in patients with prostate cancer (NCT04104607), with very favorable safety and preliminary efficacy. The optimized format that CC-3 shares with its PSMAxCD3 "sister molecule" allows for application of effective bsAb doses with expected high anticancer activity. The clinical trial comprises two phases: The first phase is a dose-escalation part to evaluate the maximally tolerated dose (MTD) of CC-3. This is followed by a dose-expansion part to defined the recommended phase II dose. A translational research program comprising, among others, analysis of CC-3 half-life and the induced immune response will serve to better define the mode of action of CC-3.

DETAILED DESCRIPTION:
Metastasized CRC is an aggressive malignant disease with poor prognosis after failure of at least three lines of previous therapy, with an accordingly high medical need for new therapeutic approaches. Except for the small population with microsatellite instability, so far no relevant progress has been achieved in CRC by immunotherapeutics. CC-3 is designed to direct T cells towards CRC tumor cells and additionally reacts with tumor vessels. If successful, the trial establishes a novel type of dual anti-cancer action by also attacking tumor blood supply and allowing for improved influx of immune effector cells and thus holds promise as a new concept of immunotherapy for cancer patients.

The rationale for the therapeutic use of CC-3 is based on its proposed mode of action as a bsAb being specifically designed to direct T cells via its CD3 binding part towards tumor target cells via its CD276 binding part. Furthermore, CC-3 also reacts with tumor vessels of CRC thereby allowing for a dual mode of anti-cancer action by also attacking tumor blood supply and allowing for improved influx of immune effector cells. Due to its unique ability to redirect T cells via CD3 for CD276 expressing tumor cell lysis, CC-3 can elicit repeated target cell elimination by cytotoxic T cells and a polyclonal response of previously primed CD4+ and CD8+ T cells. Compared to other immunotherapeutics presently being approved or in development (bsAbs with alternative formats like the authorised bsAb blinatumomab or other antibodies or CAR T cells), CC-3 is expected to offer the following major advantages:

(i) reduction of side effects due to its optimal bsAb format and choice of TAA, which will allow for application of truly effective bsAb doses and accordingly increased efficacy; (ii) CD276 enables dual targeting, thereby improving accessibility of CRC tumors to immune effector cells, as prerequisite for therapeutic success (iii) CC-3 is an "off the shelf drug" eliminating the preparative work required for CART cell generation that delays treatment; (iv) the introduction of the YTE modification will allow for prolonged half-life an thus convenient dosing scheme

Clinical trial rationale with regard to objectives and further development of CC-3

In nonclinical studies, in vitro and in vivo, proof of concept, preliminary pharmakokinetic (PK) and pharmakodynamic (PD) effects as well as toxicology have been evaluated as described in detail in the IB . However, due to differences between animal models and the human situation, some aspects have to be assessed and further characterised in humans. For example, the target mediated drug disposition (TMDD), an effect that largely influences the serum half-life of antibody molecules particularly at low concentrations, cannot be properly addressed in mice. Similar problems arise with the YTE modification, which prolongs serum half-life of antibodies in humans but not in mice.Furthermore, non-human primates (NHP) and rodents have several limitations as predictive models for toxicity and immunogenicity evaluation of CC-3. The CD3 binding part of CC-3 does not cross-react with CD3 of macaques and thus it is not possible to evaluate in these NHPs dose limiting side effects. Therefore, a First in Human clinical trial is planned for CC-3 to characterise the effects of CC-3 in humans. In general CD276 is a target antigen with particularly attractive properties. It is expressed not only on tumor cells but also on tumor vessels, allowing for "dual targeting" of a variety of solid tumors including (but not limited to) GI cancer. The importance of vascular targeting for treatment of solid tumors has been elegantly demonstrated in numerous reports.

As described in detail in the IB, CD276 is expressed on all analysed samples (n=59) of colorectal tumor samples of patients with metastazised disease. Of note, CD276 is expressed on the primary tumor as well as on metastasis. Therefore, the analysis of CD276 expression on the tumor comprises an exploratory objective of this trial but is not needed for inclusion of patients.

The phase I trial is designed to confirm and further explore the safety and tolerability of the CD276xCD3 bsAb CC-3 in adult patients with CRC after failure of at least three lines of previous therapy. The primary objectives are to define the MTD and RP2D of CC-3 and the overall safety defined as incidence and severity of AEs under therapy with CC-3. Furthermore, the trial aims to expand experience on pharmacokinetics, pharmacodynamics and toxicology of CC-3 from nonclinical- studies. A focus will be on the following specific aspects/parameters:

* PK and PD of CC-3 in humans
* Assessment of objective response rate by RECIST 1.1 on routine imaging
* Evaluatation of disease control rate (CR, PR, SD)
* Overall (OS) and progression free survival (PFS)
* Immunogenicity of CC-3 in humans based on both absolute (number and percentage of subjects who develop human anti-human antibody (HAHA).
* Overall quality of life scores (EORTC QLQ C-30)
* Absolute changes from baseline in the tumor marker (CEA und CA 19-9)
* Absolute changes from baseline in laboratory parameters
* Change in T cell activation and cytokines from baseline
* To correlate safety and efficacy of CC-3 treatment with with clinical, biological and patient characteristics
* To correlate the effect of CC-3 on serum cytokine levels and pharmarkodynamic biomarkers in the peripheral blood
* To assess long-term safety and product specific safety

Dose rationale for CC-3

Considerations on a safe starting dose of 20µg for CC-3 are, besides preclinical in vitro and in vivo data of CC-3, based on the meanwhile available PK data from a clinical study with CC-1, an identically formatted bsAb with PSMAxCD3 - (rather than CD276xCD3)-specificity, but also on clinical experience with MGD009, a bsAb with CD276xCD3-specificity as well as recently published data from several clinical studies with CD20xCD3 bsAb. The target dose of 4mg CC-3 is based on observations from the in vivo model with humanized NSG mice, where repetitive dosing with 1.4µg CC-3 was able to eradicate established flank tumors. This dose corresponds to approximately 4mg once per week in humans. Further details can be found in the IB of CC-3.

Safety and expected risks of the IMP

For CC-3, so far, no clinical safety data from other clinical trials are available. CC-3 has been preclinically characterized extensively in vitro and in vivo, the toxicity of the treatment class of bsAbs, with CRS as main class toxicity, is well known and safety data for CC-1, an identically formatted bsAb with PSMAxCD3 (rather than CD276xCD3)-specificity, which was extensively investigated in the ongoing clinical FIH study is available.

In this FIH trial (NCT04104607, DKTK_PMO_1605), investigating CC-1 in patients with CRPC, CRS was the most frequently observed toxicity, experienced by 78% of the patients. Notably, it never exceeded grade 2 after pre-emptive tocilizumab application and resolved in most cases without additional application of tocilizumab. Besides mild to moderate hypertension (observed in 50% of patients), no further CC-1 related toxicities (i.e., anaphylactic reaction) were observed. As expected and attributable to tocilizumab application, hematologic events (i.e. neutropenia, thrombocytopenia) were present in most patients, and hepatotoxicity was observed in some patients.

As CC-3 is shares the biological function with CC-1 and other bsAb, a similar or even better safety profile is expected. Especially in comparison to CC-1, with CC-3 a lower risk for CRS is expected as the CD3 binder has been attenuated. In addition, nowdays CRS is a well-known class toxicity of bsAb and risk mitigation strategies by e.g. application of tocilizumab are available. The selected dosing scheme of CC-3 in this clinical trial will not only allow for continous exposure of tumor cells to CC-3, but it is also considered to increase the tolerability of CC-3 by introduction of priming doses. Moreover, CC-3 is applied during daytime when dedicated experienced study personnel is present and can ensure close monitoring of patients during and after CC-3 application.

ELIGIBILITY:
Inclusion Criteria:

written signed informed consent

* Patient is able to understand and comply with the protocol for the duration of the clinical trial including undergoing treatment and scheduled visits and examinations
* Patients with progressing metastatic CRC who were previously treated with FOLFOX, FOLFIRI, FOLFOXIRI, TAS-102, or regorafenib, if applicable in combination with anti-VEGFR monoclonal antibody (mAb) and anti-EGFR mAb (the latter, if RAS-wild-type and left sided tumors).

In case of MSI-high/dMMR tumors, patients should have received checkpoint inhibitor therapy and at least two further lines of therapy of that stated above.

In case of patients BRAF V600E mutation patients should have received: Cetuximab in combination with encorafenib in second- or third-line treatment.

* At least one measurable lesion that can be accurately assessed at baseline by CT or MRI and is suitable for repeated assessment per RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Patient aged ≥ 18, no upper limit
* Female patients of child bearing potential (FCBP) and male patients with partners of child bearing potential, who are sexually active, must agree to the use of two effective forms (at least one highly effective method) of contraception. This should be started from the signing of the informed consent and continue throughout period of taking study treatment and for 2 months after last dose of study drug.
* For FCBP two negative pregnancy test (sensitivity of at least 25 mU/ml) prior to first application of CC-3
* All subjects must agree to refrain from donating blood while on study drug and for 2 months after last dose of CC-3.
* Adequate bone marrow, renal, and hepatic function defined by laboratory tests within 14 days prior to study treatment:

  * Hemoglobin ≥ 9 g/dl (Transfusion of packed red blood cells prior to enrolment allowed)
  * Neutrophil count ≥ 1,500/mm3
  * Platelet count ≥ 75,000/µl
  * Serum creatinine ≤ 1.5mg/dl or creatinine clearance ≥ 60ml/min
  * hepatic function of patients without current hepatic metastasis:

    * Bilirubin ≤ 1.5x upper limit of normal (ULN), in case of known Gilbert syndrome higher values are allowed if due to increase of indirect bilirubin
    * ALT and AST ≤ 2.5 x ULN
  * hepatic function of patients with current hepatic metastasis:

    * Bilirubin ≤ 2.5 x upper limit of normal (ULN)
    * ALT and AST ≤ 5. x ULN

Exclusion Criteria:

* Other malignancy requiring treatment within the last year except: adequately treated non-melanoma skin cancer and low-grade non-muscle invasive papillary bladder cancer.
* Concurrent or previous treatment within 30 days in another interventional clinical trial with an investigational anticancer therapy
* Persistent toxicity (≥ Grade 2 according to Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) caused by previous cancer therapy, excluding alopecia and neurotoxicity
* Clinical signs of active infection (> grade 2 according to CTCAE version 5.0)
* Known cerebral/meningeal manifestation of CRC
* History of HIV infection
* Viral active or chronic hepatitis (HBV or HCV)
* Ongoing autoimmune disease
* History of relevant CNS pathology or current relevant CNS pathology (e.g. seizure, paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis, coordination or movement disorder)
* Therapeutic anticoagulation therapy
* Major surgery within 4 weeks of starting study treatment. Patients must have recovered from any effects of major surgery.
* Patients receiving any systemic chemotherapy, mAb or radiotherapy within 2 (for mAb 4) weeks prior to study treatment or a longer period depending on the defined characteristics of the agents used
* Heart failure NYHA III/IV
* Severe obstructive or restrictive ventilation disorder
* Known intolerance to CC-3 or other immunoglobulin drug products as well as hypersensitivity to any of the excipients present in CC-3
* Live and live-attenuated vaccination 30 days prior to treatment
* Pregnant or breast-feeding women
* Current ileus with severely altered GI function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety 1-Adverse Events Assessment | Day 1 Day 2 Day 3 Day 8 +/- 1 day Day 9 Day 15 +/- 1 day Every 7 days +/- 2 days after Treatment week 3 7 days +/- 2 days after last CC-3 28 days +/- 2 days after last CC-3 28 days after FU +/- 3 days
  Dose escalation and dose expansion part: Characterization of the safety of CC-3 in patients with metastasized CRC, and to define the recommended phase-II dose (RP2D) of CC-3
  Adverse events should be documented and recorded continuously. Patients have to be followed for AEs from visit T1V1( treatment week1 Visit 1) up to last clinical trial visit or until all drug-related toxicities have been resolved, whichever is later, or until the investigator assesses AEs as "chronic" or "stable". Each occurrence of an AE must be reported once indicating the CTC (Version 5.0) grade. If the CTC grading of an ongoing AE changes this has to be reported. If an event stops and later restarts, all occurrences must be reported. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®) v26.0 or higher. All AEs will be graded according to the CTCAEv5.0, except for cytokine release syndrome, which will be graded according to modified criteria by Lee et al. (Lee et al., 2019).
Safety 2 -Blood Chemistry-Transaminases | Day 1 Day 2 Day 3 Day 8 +/- 1 day Day 9 Day 15 +/- 1 day Every 7 days +/- 2 days after Treatment week 3 7 days +/- 2 days after last CC-3 28 days +/- 2 days after last CC-3 28 days after FU +/- 3 days
  AST/SGOT in [U/l]
  ALT/SGPT in [U/l)
Safety 3-Hematology-haemoglobin | Day 1 Day 2 Day 3 Day 8 +/- 1 day Day 9 Day 15 +/- 1 day Every 7 days +/- 2 days after Treatment week 3 7 days +/- 2 days after last CC-3 28 days +/- 2 days after last CC-3 28 days after FU +/- 3 days
  haemoglobin in [g/l]
Safety 3-Hematology-Red Blood Cells | Day 1 Day 2 Day 3 Day 8 +/- 1 day Day 9 Day 15 +/- 1 day Every 7 days +/- 2 days after Treatment week 3 7 days +/- 2 days after last CC-3 28 days +/- 2 days after last CC-3 28 days after FU +/- 3 days
  RBC in [cells/µl]
Safety 3-Hematology-thrombocytes | Day 1 Day 2 Day 3 Day 8 +/- 1 day Day 9 Day 15 +/- 1 day Every 7 days +/- 2 days after Treatment week 3 7 days +/- 2 days after last CC-3 28 days +/- 2 days after last CC-3 28 days after FU +/- 3 days
  PLT in [cells/µl]
Safety 3-Hematology-White Blood Cells | Day 1 Day 2 Day 3 Day 8 +/- 1 day Day 9 Day 15 +/- 1 day Every 7 days +/- 2 days after Treatment week 3 7 days +/- 2 days after last CC-3 28 days +/- 2 days after last CC-3 28 days after FU +/- 3 days
  WBC in [cells/µl]

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Ott JM, Gassenmaier V, Bitzer M, Schurch CM, Heitmann JS, Hagelstein I. B7-H3: a consistent marker in metastatic colorectal cancer with potential for targeted treatment. Pathol Oncol Res. 2025 Aug 13;31:1612186. doi: 10.3389/pore.2025.1612186. eCollection 2025. PMID 40881578